CLINICAL TRIAL: NCT05573217
Title: The Utility of Cell-free DNA Methylation Markers for the Response Prediction of Systemic Treatment for Hepatocellular Carcinoma
Brief Title: The Utility of Cell-free DNA Methylation Markers for Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202106001RIPB
Record Dates: First submitted 2022-10-03; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Cell-free Methylation Markers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The subjects of this study were patients with liver cancer diagnosed by physicians according to AASLD clinical criteria or pathological biopsy.

Those who plan to receive systemic drug treatment for liver cancer in National Taiwan University Hospital include Nexavar, Lenvatinib, Avastin, Tecentriq, Strivarga, Cabometyx, Cyramza, Nivolunab, Pembrolizumab, and Yervoy. Weak and uncooperative patients were excluded from blood tests, which were performed with full informed consent for relevant tumor markers (AFP ,PIVKA-II and methylation analysis). The data are then counted and compared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with liver cancer by AASLD clinical criteria or pathological slides Patients planning to receive systemic drug therapy for liver cancer at National Taiwan University Hospital include Nexavar, Lenvatinib, Avastin, Tecentriq, Strivarga, Cabometyx, Cyramza, Nivolunab, Pembrolizumab, and Yevoy.
2. Over 20 years old.
3. In the case of informed consent, willing to sign the consent form of the subjects.

Exclusion Criteria:

1. Patients who are weak and unable to cooperate with blood test.
2. Kidney dysfunction, serum creatinine greater than 1.5 x UNL (normal value) and no hemodialysis treatment, who are judged to be unwell for computed tomography or MRI contrast agent injection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with liver cancer by AASLD clinical criteria or pathological slides Patients planning to receive systemic drug therapy for liver cancer at National Taiwan University Hospital include Nexavar, Lenvatinib, Avastin, Tecentriq, Strivarga, Cabometyx, Cyramza, Nivolunab, Pembrolizumab, and Yevoy.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate efficacy | 3 month after treatment
  Correlation of methylation profiling results and tumor treatment response.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No